CLINICAL TRIAL: NCT06299735
Title: Comparison of Postoperative Pulmonary Complications in Patients Undergoing Minimal Invasive Cardiac Surgeries With the Use of Bronchial Blocker and Double-Lumen Tube in Airway Management
Brief Title: Comparison of Airway Management With Bronchial Blocker and Double-Lumen Tube in Single-Lung Ventilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AsenaIremYildiz1
Record Dates: First submitted 2024-02-06; First posted 2024-03-08 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Heart Valvular Disease; Coronary Arteriosclerosis; One-lung Ventilation
Keywords: postoperative pulmonary complications; minimally invasive cardiac surgery; one lung ventilation
MeSH Terms: conditions — Heart Valve Diseases; Coronary Artery Disease | interventions — Airway Management

STUDY DESIGN:
Intervention Model Description: The anesthesia method applied for both patient groups is the same. However, the airway maintenance device used will vary between two different patient groups. Group BB: A bronchial blocker will be used for this patient group, Group DLT: A double-lumen tube will be used for this patient group. The parameters to be recorded for both patient groups include: preoperative smoking history, ARISCAT score, systolic arterial pressure, diastolic arterial pressure, saturation, pulse, and the duration of airway device insertion following anesthesia induction and intubation. For the assessment of postoperative pulmonary complications in both patient groups, arterial blood gas analysis, chest X-ray, respiratory sounds, and the patient's oxygen requirement will be monitored every 6 hours for 24 hours.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group using a double-lumen tube for single-lung ventilation (Active Comparator): Group DLT: For the assessment of postoperative pulmonary complications, arterial blood gas analysis, chest X-ray, respiratory sounds, and the patient's oxygen requirement will be monitored every 6 hours for 24 hours. The parameters to be examined preoperatively are: smoking history, ARISCAT score (Age, Preoperative SpO₂, Respiratory infection in the last month, Preoperative anemia (Hgb ≤10 g/dL), Surgical incision, Duration of surgery, Emergency procedure).
  Interventions: Procedure: Minimally Invasive Cardiac Surgery (airway management with double-lumen tube)
- Patient group using a endobronchial blocker for single-lung ventilation (Active Comparator): Group BB: For the assessment of postoperative pulmonary complications, arterial blood gas analysis, chest X-ray, respiratory sounds, and the patient's oxygen requirement will be monitored every 6 hours for 24 hours. The parameters to be examined preoperatively are: smoking history, ARISCAT score (Age, Preoperative SpO₂, Respiratory infection in the last month, Preoperative anemia (Hgb ≤10 g/dL), Surgical incision, Duration of surgery, Emergency procedure).
  Interventions: Procedure: Minimally Invasive Cardiac Surgery (airway management with endobronchial blocker)

INTERVENTIONS:
Procedure: Minimally Invasive Cardiac Surgery (airway management with double-lumen tube) — Anesthesia induction will involve 1 mg/kg lidocaine, 1 µg/kg fentanyl, 1 mg/kg propofol, and 0.7 mg/kg rocuronium. Following anesthesia induction, a double-lumen tube will be inserted.Subsequently, patients will be connected to a mechanical ventilator. Tube placement will be confirmed using fiberoptic bronchoscopy.
  Arms: Patient group using a double-lumen tube for single-lung ventilation
Procedure: Minimally Invasive Cardiac Surgery (airway management with endobronchial blocker) — Anesthesia induction will involve 1 mg/kg lidocaine, 1 µg/kg fentanyl, 1 mg/kg propofol, and 0.7 mg/kg rocuronium. Following anesthesia induction, endotracheal tube-bronchial blocker will be inserted.Subsequently, patients will be connected to a mechanical ventilator. Tube placement will be confirmed using fiberoptic bronchoscopy.
  Arms: Patient group using a endobronchial blocker for single-lung ventilation

SUMMARY:
In this study, the primary aim is to compare the impact of using a double-lumen tube and bronchial blocker for single-lung ventilation in patients undergoing minimal invasive cardiac surgeries on postoperative pulmonary functions. Secondary objectives include the comparison of application duration, success in lung collapse, and the number of repositioning attempts for both techniques.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized clinical trial. After obtaining ethical approval, 66 patients meeting the inclusion criteria and providing consent, who will undergo minimal invasive cardiac surgery at Ankara City Hospital Heart and Vascular Hospital Operating Room, will be included in the study. Patients will be randomized into two groups using a sealed envelope method (Group DLT: Group undergoing Single-Lung Ventilation with a Double-Lumen Tube, and Group BB: Group undergoing Single-Lung Ventilation with a bronchial blocker within a single-lumen Endotracheal Tube). Both groups will receive standard anesthesia induction and maintenance. Patients brought to the operating room without premedication will start invasive blood pressure monitoring with awake intra-arterial cannulation in addition to standard ASA monitoring.

Anesthesia induction will be performed with 1 mg/kg lidocaine, 1 µg/kg fentanyl, 1 mg/kg propofol, and 0.7 mg/kg rocuronium. After 3 minutes of anesthesia induction, a double-lumen tube/endotracheal tube-bronchial blocker of the appropriate size based on patients' height and gender will be placed. Tube placement will be confirmed with the assistance of a flexible bronchoscope in both groups. During anesthesia maintenance, the gas mixture of 50%/50% oxygen/air with 1-2% sevoflurane will be adjusted to maintain BIS between 40-60. During mechanical ventilation, in both groups, tidal volume of 6-8 ml/kg, respiratory rate of 10-12/min, and PEEP of 4-5 cmH2O will be set for double-lung ventilation, and for single-lung ventilation, tidal volume of 4-6 ml/kg, respiratory rate of 12-14/min, and PEEP of 4-5 cmH2O will be adjusted to maintain PIP<25cmH2O, SpO2>90, and PaCO2<40 mmHg (based on ideal body weight).

Apart from the two compared airway management techniques, both groups will receive standard anesthetic care, multimodal analgesia, and cardiopulmonary bypass method. Determining the impact of these methods on pulmonary functions is crucial to avoid adding potential pulmonary complications related to the inflammatory damage caused by the cardiopulmonary bypass pump to the airway management used for single-lung ventilation. Additionally, comparing the rates of technical complications and placement times for these techniques can guide anesthesia management. Both techniques are routinely used in our clinic for the minimal invasive cardiac surgery procedure based on the preference of anesthesia providers.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for on-pump minimal invasive cardiac surgical procedures requiring single-lung ventilation
* Female and male patients aged 18 and above
* Patients with ASA scores of 1-2-3
* Patients with signed informed consent to participate in the study
* Patients with a Body Mass Index (BMI) less than 40

Exclusion Criteria:

* Emergency surgeries
* Patients with ASA scores greater than 3
* Advanced-stage organ (heart, kidney, liver, lung) failure
* Advanced lung diseases (COPD, FEV1<50%, restrictive lung diseases, history of chest surgery, Pulmonary Hypertension, PAB>30mmHg)
* Patients with anticipated difficult intubation
* Pregnant individuals
* Patients with a BMI greater than 40
* Patients lacking the ability to read, understand, sign the informed consent form, and those who do not wish to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of Postoperative Pulmonary Complications in Patient Groups Undergoing Single-Lung Ventilation with Double-Lumen Tube and Bronchial Blocker | Postoperative 7 days
  Until discharge;
  * Patients will be regularly visited during the postoperative period.
  * Arterial blood gas analysis will be conducted at 6-hour intervals within the first 24 hours, and if necessary thereafter.
  * Respiratory sounds will be auscultated daily.
  * Chest X-rays will be taken every day.
  The presence of pneumothorax, atelectasis, hemothorax, pneumonia, or ARDS in patients will be observed and recorded.

SECONDARY OUTCOMES:
Duration of insertion of the double-lumen tube / bronchial blocker | 30 minutes
  In Double Lumen Tube group : The time elapsed from the beginning of laryngoscopy following the induction of general anesthesia to the placement of the double-lumen tube and its confirmation with fiberoptic bronchoscopy.
  In Bronchial Blocker group : The time elapsed from the beginning of laryngoscopy following the induction of general anesthesia to the completion of endotracheal tube placement, and subsequently, the placement of the bronchial blocker under fiberoptic bronchoscopy guidance will be recorded.
Incidence of postoperative sore throat | Postoperative 7 days
  Patients will be visited daily during the postoperative period, and they will be asked if they have sore throat . The intensity of throat pain will be assessed using a visual analog scale. Patients will be asked to assign a number from 0 to 10 to describe the severity of their pain (0: no pain, 10: severe pain ) and it will be recorded.
Incidence of postoperative hoarseness | Postoperative 7 days
  Patients will be visited daily during the postoperative period, and they will be asked if they have hoarseness and it will be recorded as either yes or no.
Impact of the success of lung collapse | Until the end of the operation (maximum 12 hours )
  End of the surgery, the surgeon will be asked about the level of lung collapse, and they will be requested to assign a number indicating the level of maximum collapse on a verbal rating scale from 0 to 10. (0 :no lung collapse, 10: complete collapse) And it will be recorded.
Satisfactory lung collapse time | Until the end of the operation (maximum 12 hours )
  After one lung ventilation begins, the surgeon will be asked about the level of lung collapse,and they will be instructed to notify when satisfactory lung collapse (when the collapse score of 8) is achieved.The time elapsed from the initiation of single-lung ventilation until satisfactory collapse is achieved will be recorded. ( minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Nevriye Salman, Principal Investigator — ankara bilkent city hospital, anesthesiology and reanimation clinic
Locations (1):
- Ankara bilkent city hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ganapathy S. Anaesthesia for minimally invasive cardiac surgery. Best Pract Res Clin Anaesthesiol. 2002 Mar;16(1):63-80. doi: 10.1053/bean.2001.0208. PMID 12491544
- [Result] Vernick W, Atluri P. Robotic and minimally invasive cardiac surgery. Anesthesiol Clin. 2013 Jun;31(2):299-320. doi: 10.1016/j.anclin.2012.12.002. Epub 2013 Mar 13. PMID 23711646
- [Result] Patel M, Wilson A, Ong C. Double-lumen tubes and bronchial blockers. BJA Educ. 2023 Nov;23(11):416-424. doi: 10.1016/j.bjae.2023.07.001. Epub 2023 Sep 18. No abstract available. PMID 37876764
- [Result] Knoll H, Ziegeler S, Schreiber JU, Buchinger H, Bialas P, Semyonov K, Graeter T, Mencke T. Airway injuries after one-lung ventilation: a comparison between double-lumen tube and endobronchial blocker: a randomized, prospective, controlled trial. Anesthesiology. 2006 Sep;105(3):471-7. doi: 10.1097/00000542-200609000-00009. PMID 16931978
- [Result] Kottenberg-Assenmacher E, Kamler M, Peters J. Minimally invasive endoscopic port-access intracardiac surgery with one lung ventilation: impact on gas exchange and anaesthesia resources. Anaesthesia. 2007 Mar;62(3):231-8. doi: 10.1111/j.1365-2044.2007.04954.x. PMID 17300299
- [Result] Ender J, Bury AM, Raumanns J, Schlunken S, Kiefer H, Bellinghausen W, Petry A. The use of a bronchial blocker compared with a double-lumen tube for single-lung ventilation during minimally invasive direct coronary artery bypass surgery. J Cardiothorac Vasc Anesth. 2002 Aug;16(4):452-5. doi: 10.1053/jcan.2002.125144. PMID 12154424
- [Result] Ko R, McRae K, Darling G, Waddell TK, McGlade D, Cheung K, Katz J, Slinger P. The use of air in the inspired gas mixture during two-lung ventilation delays lung collapse during one-lung ventilation. Anesth Analg. 2009 Apr;108(4):1092-6. doi: 10.1213/ane.0b013e318195415f. PMID 19299766
- [Result] Zhang Y, Yan W, Fan Z, Kang X, Tan H, Fu H, Li Z, Chen KN, Chen J. Preemptive one lung ventilation enhances lung collapse during thoracoscopic surgery: A randomized controlled trial. Thorac Cancer. 2019 Jun;10(6):1448-1452. doi: 10.1111/1759-7714.13091. Epub 2019 May 21. PMID 31115153